CLINICAL TRIAL: NCT00680732
Title: Prevention of Intrauterine Growth Retardation in Hounde District, Burkina Faso: the Malaria Component
Brief Title: Prevention of Intrauterine Growth Retardation in Burkina Faso: the Malaria Component
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Departments of Parasitology and Public Health, ITM, Antwerp, Belgium (Unknown); Centre Muraz (Other); Laboratoire National de Santé Publique, Ouagadougou, Burkina Faso (Unknown)
Responsible Party: Prof. Umberto D'Alessandro, Head of the Parasitology Department, ITM
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IUGR Malaria
Record Dates: First submitted 2008-04-23; First posted 2008-05-20 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Malaria; Malaria in Pregnancy
Keywords: Malaria; Pregnancy; Prevention; Chloroquine; Sulphadoxine pyrimethamine; Maternal anaemia; Birth weight; Foetal anaemia
MeSH Terms: conditions — Malaria; Birth Weight | interventions — Iron; Folic Acid; Chloroquine; fanasil, pyrimethamine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A1 (Experimental): Multiple micronutrients supplements (MMS) and weekly chloroquine (CQ)
  Interventions: Dietary Supplement: Multiple micronutrients supplements (MMS); Drug: Chloroquine (CQ)
- A2 (Experimental): Multiple micronutrients supplements (MMS) and intermittent suplphadoxyne-pyrimethamine (SP)
  Interventions: Dietary Supplement: Multiple micronutrients supplements (MMS); Drug: Sulphadoxyne-pyrimethamine (SP)
- B1 (Experimental): Iron and folic acid (IFA) and weekly chloroquine (CQ)
  Interventions: Dietary Supplement: Iron and folic acid (IFA); Drug: Chloroquine (CQ)
- B2 (Experimental): Iron and folic acid (IFA) and intermittent sulphadoxyne-pyrimethamine (SP)
  Interventions: Dietary Supplement: Iron and folic acid (IFA); Drug: Sulphadoxyne-pyrimethamine (SP)

INTERVENTIONS:
Dietary Supplement: Multiple micronutrients supplements (MMS) — Vitamin A 800 mcg; vitamin E 10 mg; vitamin D 5 mcg; vitamin B1 1.4 mg; vitamin B2 1.4 mg;niacin 18 mg; vitamin B6 1.9 mg; vitamin B12 2.6 mcg; folic acid 400 mcg; vitamin C 70 mg; iron 30 mg; zinc 15 mg; copper 2 mg; selenium 65 mcg; iodine 150 mcg
  Other Names: UNIMMAP
  Arms: A1; A2
Dietary Supplement: Iron and folic acid (IFA) — Iron 60 mg and folic acid 400 mcg
  Arms: B1; B2
Drug: Chloroquine (CQ) — Tablets 100 mg of chloroquine base
  Arms: A1; B1
Drug: Sulphadoxyne-pyrimethamine (SP) — Tablets
  Other Names: Fansidar
  Arms: A2; B2

SUMMARY:
Our objective was to investigate the importance of malaria infection/disease during pregnancy and more particularly during the first trimester; we also looked at the maternal-foetal interactions and their influence on the subsequent child's response to malaria infections during the first year of life. This study was carried out !in the same population recruited for the IUGR study (NCT00642408).

DETAILED DESCRIPTION:
A research project aiming at investigating the impact of multivitamin-mineral supplementation (MMS) during pregnancy on intra-uterin growth retardation was carried out in the Hounde district, an area not far from the Centre Muraz located in Bobo Dioulasso, and where malaria is endemic. Malaria during pregnancy increases the risk of low birth weight, infant mortality and morbidity during the first year of life by inducing growth retardation, prematurity and infant anaemia.

The administration of an antimalarial drug during pregnancy has a beneficial effect on the mother and child's health by preventing malaria infection and its consequences. However, most studies have been carried out during the second or third trimester of pregnancy: the effect of malaria infection during the first trimester on the mother's and child's health is unknown. It has been reported that even one single infection may have a significant impact on the outcome of pregnancy: if it is true, then early chemoprophylaxis may have an additional advantage.

An alternative approach is the administration of intermittent presumptive treatment, which may achieve equal efficacy to continuos chemoprophylaxis; however, no studies compared effective weekly malaria chemoprophylaxis with effective intermittent presumptive treatment. Moreover, the incidence of malaria clinical episodes during SP intermittent preventive treatment has never been investigated.

Therefore, this open label, factorial study was carried out in the same women recruited for the IUGR nutritional study (NCT00642408). Women receiving multiple micronutrients supplements (MMS) or dietary supplements (IFA) were further randomised in 2 groups: CQ weekly chemoprophylaxis or SP intermittent preventive treatment. The administration of treatment was directly observed.

ELIGIBILITY:
Inclusion Criteria:

* 15 to 44 years
* females
* living in the study area

Exclusion Criteria:

* planning to move outside the district within two years
* regularly using a contraceptive methods
* already pregnant at the start of the trial

Ages: 15 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1370 (Actual)
Dates: Start 2003-06; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of standard antimalarial treatment in preventing clinical malaria in pregnant women under weekly chemoprophylaxis or intermittent treatment. | Up to delivery

SECONDARY OUTCOMES:
To determine if the occurrence of malaria during pregnancy influences the incidence of clinical malaria in infants during their first year of life. | Up to one year after delivery
To determine the burden of clinical malaria during pregnancy and its consequences on maternal anaemia, new birth weight and foetal anaemia. | Up to delivery
Effect of standard antimalarial treatment on the selection of resistant parasites in pregnant women under weekly chemoprophylaxis or intermittent treatment. | Up to one year after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Marie Claire Henry, MD, Principal Investigator — Centre Muraz
Locations (1):
- Centre Muraz, Bobo-Dioulasso, Burkina Faso